CLINICAL TRIAL: NCT02348697
Title: Non-Interventional Study to Evaluate Safety and Efficacy of NOVOCART 3D in Patients With Cartilage Defects
Acronym: NISANIK
Status: Completed | Type: Observational
Sponsor: Tetec AG (Industry)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1418; 2015-000166-62 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-28 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-01

CONDITIONS: Cartilage Diseases
Keywords: Cartilage Defect in the Knee; MACT
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: NOVOCART 3D — Autologous Chondrocyte Implantation

SUMMARY:
Non-interventional study to evaluate safety and efficacy of NOVOCART 3D in adult and adolescent patients with full thickness cartilage defects after the treatment with NOVOCART 3D.

DETAILED DESCRIPTION:
A 36-month post treatment follow up of adverse and serious adverse effects as well as the measurement of efficacy with the International Knee Documentation Committee (IKDC) Score.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients
* Children and adolescents with closed epiphysial plate
* Defect size ≥2.5 and ≤10 cm2 post-debridement
* Localized full thickness articular cartilage defect of the knee (Grade 3 & 4 International Cartilage Repair Society (ICRS) classification)

Exclusion Criteria:

* Radiologically apparent degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade >2
* More than 2 defects or 2 corresponding lesions
* Ankylosis
* Arthrofibrosis
* Diffuse chondromalacia
* Total/subtotal resected meniscus
* Insufficient Ligament guidance
* Patella malignement
* Inflammatory joint disease
* General cartilage degeneration or increased joint deterioration
* Cancer, present or within the last 5 years
* Primary treatment in children and adolescents with open epiphysial plate
* Chronical infection diseases
* Untreated coagulation disorder
* Pregnancy and lactating
* Known history of allergies against ingredients of NOVOCART® 3D

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: specialist clinical centre
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Safety - Number of Adverse Drug Reaction/Serious Adverse Drug Reaction as a Measure of Safety | 36 month
  Number of Adverse Drug Reaction/Serious Adverse Drug Reaction as a Measure of Safety

SECONDARY OUTCOMES:
Efficacy - International Knee Documentation Committee (IKDC) 2000 | 36 month
  International Knee Documentation Committee (IKDC) 2000

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kirner, PhD, Study Director — TETEC AG Reutlingen
Locations (9):
- Germany (9):
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Bamberg
  - Gelenk Klinik Orthopaedic Clinic, Gundelfingen
  - Diakoniekrankenhaus Henriettenstiftung gGmbH, Hanover
  - Heidelberg University Hospital, Heidelberg
  - Lubinus Clinicum, Kiel
  - Theresienkrankenhaus, Mannheim
  - Department of Orthopedic Surgery and the Department of Physical Medicine and Rehabilitation LMU Munich, Munich
  - Klinik rechts der Isar, München
  - University Hospital Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No